CLINICAL TRIAL: NCT07148947
Title: A Phase 2 Trial Investigating the Addition of Pacritinib to a Hypomethylating Agent as a Bridge to Allogeneic Hematopoietic Stem Cell Transplant in Patients With Accelerated and Blast Phase Myeloproliferative Neoplasms
Brief Title: Pacritinib With Standard of Care Azacitidine or Decitabine as a Bridge to Allogeneic Hematopoietic Stem Cell Transplant for Patients With Accelerated and Blast Phase Myeloproliferative Neoplasms
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125470; NCI-2025-05720 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0021044 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Accelerated Phase Myeloproliferative Neoplasm; Blast Phase Myeloproliferative Neoplasm
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Decitabine; Injections; decitabine and cedazuridine drug combination; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pacritinib and HMA bridge therapy) (Experimental): Patients receive pacritinib PO BID on days 1-28 of each cycle, starting 7 days before or 30 days after standard of care HMA bridge therapy. Cycles repeat every 28 days for 6 cycles. Patients receive HMA bridge therapy per treating physician's standard institutional practice with azacitidine IV or SC, or decitabine IV or cedazuridine/decitabine PO per standard of care. Treatment is given in the absence of unacceptable toxicity. Patents also undergo bone marrow aspiration and/or biopsy and blood sample collection during screening and as clinically indicated throughout the study.
  Interventions: Drug: Pacritinib; Drug: Decitabine; Drug: Decitabine and Cedazuridine; Drug: Azacitidine; Other: Survey Administration; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Drug: Pacritinib — Given PO
  Other Names: Oral JAK2 Inhibitor SB1518; SB 1518; SB-1518; SB1518
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Survey Administration — Ancillary studies
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy

SUMMARY:
This phase II trial tests if adding pacritinib to standard of care azacitidine or decitabine increases the number of patients able to proceed to hematopoietic stem cell transplantation (bridging) for patients with accelerated and blast phase myeloproliferative neoplasms. Pacritinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Azacitidine and decitabine are in a class of medications called hypomethylation agents. They work by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Adding pacritinib to standard of care azacitidine or decitabine may increase the number of patients able to proceed to hematopoietic stem cell transplantation for patients with accelerated and blast phase myeloproliferative neoplasms.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pacritinib orally (PO) twice daily (BID) on days 1-28 of each cycle, starting 7 days before or 30 days after standard of care hypomethylating agent (HMA) bridge therapy. Cycles repeat every 28 days for 6 cycles. Patients receive HMA bridge therapy per treating physician's standard institutional practice with azacitidine intravenously (IV) or subcutaneously (SC), or decitabine IV or cedazuridine/decitabine PO per standard of care. Treatment is given in the absence of unacceptable toxicity. Patents also undergo bone marrow aspiration and/or biopsy and blood sample collection during screening and as clinically indicated throughout the study.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* History of myeloproliferative neoplasms (MPN) as defined by the 2016 and 2022 World Health Organization criteria, with now pathologically confirmed ≥ 5% blasts in the bone marrow or peripheral blood. Prior MPNs could include polycythemia vera, essential thrombocythemia, primary myelofibrosis, secondary myelofibrosis, MPN-unclassifiable, and myelodysplastic syndrome (MDS)/MPN overlap syndromes
* Outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution by pathology. Flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 OR Karnofsky ≥ 60%
* Serum creatinine clearance ≥ 50 ml/min calculated by the Cockcroft-Gault Equation (assessed within 14 days of study day 1)
* Total bilirubin ≤ 3 (total bilirubin > 3 is allowable if thought due to Gilbert's disease, hemolysis, or MPN disease) (assessed within 14 days of study day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x upper limits of normal (ULN) (total bilirubin > 3 is allowable if thought due to Gilbert's disease, hemolysis, or MPN disease) (assessed within 14 days of study day 1)
* Patient is considered a potential transplant candidate. The attending/treating physician will determine transplant candidacy at the time of consent
* Intention to initiate therapy with an HMA per treating physician's standard institutional practice. Allowable HMAs include:

  * Azacitidine given IV or SC
  * Decitabine given IV, and
  * Decitabine given orally (as Inqovi [cedazuridine/decitabine]). If the HMA was already initiated, patients must be registered and start pacritinib within 30 days of initiation
* Hyperleukocytosis, white blood cell (WBC) > 100,000/μL, or with concern for other complications of high tumor burden or leukostasis (e.g. hypoxia, disseminated intravascular coagulation) can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) any time prior to enrollment
* Women of child-bearing potential and men must be agree to use a highly effective method of contraception, starting at the first dose of study therapy through 90 days after the last dose of study therapy
* Capable of providing valid informed consent

Exclusion Criteria:

* Previous treatment with chemotherapy (e.g. hypomethylating agents or cytarabine-based regimens) for MPN (does not include the first cycle of treatment with an allowable HMA initiated within 30 days prior to start of pacritinib). Prior temporary measures to control blood counts is allowed. Prior treatment with hydroxyurea, interferons or JAK inhibitor therapy (including pacritinib) is allowed
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, HIV])
* Known hypersensitivity to any study drug
* Females who are pregnant or breastfeeding (Women of childbearing potential [WOCBP] must have a negative serum pregnancy test within 14 days prior to enrollment)
* Treatment with any other anti-MDS/leukemia investigational agent within 2 weeks of start of study drugs
* Corrected QT interval (QTC) > 480 msec as measured by the Fridericia formula (changing of medications/supplementing electrolytes is allowed to determine if this helps QTc reduce to < 480 msec)
* Concurrent use of a strong CYP3A4 inhibitor or inducer at enrollment that cannot be discontinued (washout period ≥ 5 half-lives prior to day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who receive hematopoietic stem cell transplant | Up to 9 months from starting treatment
  Will be estimated and reported with a 95% confidence interval using methodology to account for the two-stage design.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No